CLINICAL TRIAL: NCT00941642
Title: Placebo Controlled Study Using Lovaza as Treatment for Non-Alcoholic Fatty Liver Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huntington Medical Research Institutes (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Edward A. Mena, MD, Huntington Medical Research Institutes
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: LOVAZA - NAFLD; IND # 105,085.
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Nonalcoholic Fatty Liver Disease (NAFLD); Lovaza; Steatosis; Non-Alcoholic steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lovaza (Active Comparator): Single blind, active treatment arm Lovaza, is the only fish oil supplement approved by the FDA. The Lovaza treatment group will take 4g of Lovaza daily for a minimum of 48 weeks.
  Interventions: Drug: Lovaza
- Placebo (Placebo Comparator): Single blind, Placebo arm study drug will contain 994.0 mg of corn oil and 6mg of alpha tocopherol as an excipient in a soft gelatin capsule shell. Subjects will take 4g daily for a minimum of 48 weeks.
  Interventions: Drug: placebo control

INTERVENTIONS:
Drug: Lovaza — Approximately 50% of study subjects will be randomized to the active treatment arm -Lovaza. Subjects will be dosed with 4g of Lovaza gel capsules daily for a minimum of 48 weeks duration.
  Arms: Lovaza
Drug: placebo control — Approximately 50% of study subjects will be randomized to the placebo arm of this study. Placebo arm subjects will receive 4g of placebo gel caps daily for a minimum of 48 weeks duration.
  Arms: Placebo

SUMMARY:
Lovaza is the only fish oil supplement approved by the FDA. It is available by prescription for the treatment of hypertriglyceridemia (> 500 mg/dl). The primary mechanism appears to be a reduction in hepatic production of triglycerides. Also decreases the hepatic production of very low density lipoprotein (VLDL). There also may be antioxidant properties as well. The thought behind using Lovaza as a treatment for non-alcoholic fatty liver disease (NAFLD) is two fold. It would help in the decrease production of triglycerides by the liver and have antioxidant properties decreasing the production of free radicals in the liver. In doing so, steatohepatitis, fibrosis, and perhaps cirrhosis and liver cancer would be prevented.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Abnormal liver enzymes >40 IU/L. Definition of normal is ALT 19 for a woman and 30 for a man.
* Patients must meet ATP III criteria for metabolic syndrome: Central obesity as measured by waist circumference. Men - greater than or equal to 40 inches. Women - greater than or equal to 35 inches.
* Blood HDL cholesterol. Men - less than 40 mg/dL. Women - less than 50 mg /dL.
* Blood pressure greater than or equal to 130/85.
* Fasting glucose greater than or equal to 100 mg/dL but less than 126mg/dL on 2 separate occasions.
* Fasting blood triglycerides greater than or equal to 150 mg/dL.
* Hepatitis B and C negative
* Autoimmune Hepatitis, Wilson's Disease, Hemochromatosis negative, etc.
* NASH or NAFLD on biopsy of any degree:

Exclusion Criteria:

* Below the age of 18.
* Other Causes of Liver inflammation.
* Daily alcohol consumption in excess of 20 grams / day for men and 10 grams / day for women. If participant unable to quantify his/her alcohol intake, they should be excluded.
* Taking a prescribed medication know to cause fatty liver disease 6 months prior to enrollment. Also, subjects with secondary causes of fatty liver disease (ie. Gastric bypass) should be excluded from the study.
* Cirrhosis.
* Subjects on oral insulin-sensitizing agents and other drugs currently being used in the treatment of NAFLD. Such agents include fibrates, Vitamin E, S-adenosyl-methionine, betaine, N-acetylcysteine, and milk thistle extracts.
* Diabetes (fasting sugar above 126mg/dl).
* Pregnancy or lactation. Women of child bearing potential must have a negative serum pregnancy test at screening, a negative urine pregnancy test prior to treatment and be practicing an acceptable form of barrier contraception for the duration of the study.
* Any serious or chronic disease that in the opinion of the Principal Investigator (PI), may affect the assessment of safety or efficacy parameters. This includes but is not limited to, patients with malignancy, other than Basal Cell Carcinomas.
* Patients who, in the opinion of the site PI, are not suitable candidates for enrollment or would not comply with the requirements of the study.
* Patients who have had a liver transplant.
* Any allergy to fish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
To determine if Lovaza improves fibrosis and the NASH activity index. | 48 weeks

SECONDARY OUTCOMES:
To determine if Lovaza improves AST/ALT level and improves steatosis on biopsy. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Mena, MD, Principal Investigator — Huntington Medical Research Institutes - Liver Center; Myron J Tong, PhD, MD., Study Director — Huntington Medical Research Institutes - Liver Center
Locations (1):
- HMRI - Liver Center, Pasadena, California, United States